CLINICAL TRIAL: NCT05144724
Title: Volume Targeted Mask Ventilation Versus Pressure Ventilation in Preterm Infants
Acronym: VOLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00115050
Record Dates: First submitted 2021-10-21; First posted 2021-12-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Respiratory Distress
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volume Targeted Ventilation (Experimental): Positive pressure ventilation will be provided using a set tidal volume
  Interventions: Procedure: Volume targeted ventilation
- Pressure guided Ventilation (Active Comparator): Positive pressure ventilation will be provided using a set peak inflation pressure
  Interventions: Procedure: Pressure targeted ventilation

INTERVENTIONS:
Procedure: Volume targeted ventilation — Positive pressure ventilation will be provided using a set tidal volume
  Arms: Volume Targeted Ventilation
Procedure: Pressure targeted ventilation — Positive pressure ventilation will be provided using a set peak inflation pressure
  Arms: Pressure guided Ventilation

SUMMARY:
This is a pilot trial to assess the feasibility of volume Targeted Ventilation in the Delivery Room.

Preterm infants will be randomized to pressure guided or volume targeted ventilation during respiratory support in the delivery room

ELIGIBILITY:
Inclusion Criteria:

* Born between 23+0/7 to 28+6/7 weeks' gestation
* Considered suitable for full resuscitation, i.e., no parental request or antenatal decision to forego resuscitation
* Informed parental consent

Exclusion Criteria:

* Major congenital or chromosomal malformation
* Conditions that might have an adverse effect on breathing or ventilation (e.g., high risk for lung hypoplasia, congenital diaphragmatic hernia)
* Congenital heart disease requiring intervention in the neonatal period
* Hydrops requiring intervention in the neonatal period
* Neonatal resuscitation initiated before NICU team arrival
* Infants who are born outside of study center and transported to center after delivery

Ages: 0 Minutes to 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Percentage of of eligible participants (=infants requiring PPV) who have the intervention performed correctly without protocol deviation (=cross over to control group when randomized to VTV-group) | Through study completion (total 18 months)
  Percentage of Participants who have received allocated treatment

SECONDARY OUTCOMES:
Number of participants with mortality | up to 6 months of NICU admission
  Infants who died during NICU admission - all-cause in-hospital
Number of participants with severe brain injury on cranial ultrasound | up to 6 months of NICU admission
  Severe grade 3 and 4 intraventricular or intraparenchymal hemorrhage according to Papile, periventricular leukomalacia, or ventriculomegaly based on neuroimaging studies (timing and frequency of imaging based on local site practices)
Number of participants with severe retinopathy of prematurity (stage 3 or higher) | up to 6 months of NICU admission
  Defined in the International Classification of ROP, and/or ROP treated with laser, cryotherapy, or intraocular injection therap
Number of participants with bronchopulmonary dysplasia at 36 weeks corrected age | At 36 weeks corrected age
  Defined as receiving any supplemental oxygen or any form of respiratory support (including invasive mechanical ventilation, non-invasive ventilation with continuous positive airway pressure, nasal intermittent positive pressure ventilation, or high-flow nasal canula)
Number of participants with Bronchopulmonary dysplasia at 40 weeks corrected age | At 40 weeks corrected age
  Defined as receiving any supplemental oxygen or any form of respiratory support (including invasive mechanical ventilation, non-invasive ventilation with continuous positive airway pressure, nasal intermittent positive pressure ventilation, or high-flow nasal canula)
Total duration of mechanical ventilation via an endotracheal tube in days | Days during NICU admission (up to 6 months)
  Count of days in were an endotracheal tube was placed and the infant was mechanical ventilation
Number of participants discharge home on oxygen | At time of NICU discharge (with 6 moths from birth)
  Infants being discharged home with oxygen
Duration of any respiratory support in days | Days during NICU admission (up to 6 months)
  Defined as invasive mechanical ventilation, non-invasive ventilation with continuous positive airway pressure, nasal intermittent positive pressure ventilation, or non-invasive neural assist ventilation or non-invasive high frequency ventilation, or high-flow nasal cannula) in days
Duration of supplemental oxygen in days | Days during NICU admission (up to 6 months)
  Count of days in were the infant received supplemental oxygen
Length of hospital stay in days | Number of days from birth to discharge (up to 6 months)
  Defined as number of days from birth to discharge
Rate of intubation in the delivery room | within 60min after birth
  Infants who were intubated in the delivery room at birth
Rate of chest compression in the delivery room | within 60min after birth
  Infants who received chest compression in the delivery room at birth
Rate of pneumothorax | up to 6 months of NICU admission
  Diagnosed by chest x-ray or lung ultrasound) and interventions (e.g., needle drainage or chest drain)
Number of participants with necrotizing enterocolitis | up to 6 months of NICU admission
  Defined as modified Bell's criteria stage 2 or greater
Duration of positive pressure ventilation at birth in days | within the first 10 min after birth
  Infants who received positive pressure ventilation in the delivery room at birth

OTHER OUTCOMES:
Resuscitators subjective workload performing mask ventilation | within the first 10 min after birth
  Es evaluated by Surgery Task Load Index (SURG-TLX)-questionnaire.
Resuscitators qualitative feedback on using VTV-PPV in the delivery room | within the first 10 min after birth
  Provided through free text responses

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmölzer, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
The protocol will be published in an open access journal and data can be requested from the principal investigator
Supporting Information: Study Protocol, ICF
Time Frame: Protocol will be published within 18 months

REFERENCES:
- [Derived] Law BHY, Yaskina M, Davis PG, Polglase G, Dunn M, Mukerji A, Schmolzer GM. Study protocol for the volume targeted mask ventilation versus pressure ventilation in preterm infants-the VOLT-trial. Front Pediatr. 2026 Jan 6;13:1743460. doi: 10.3389/fped.2025.1743460. eCollection 2025. PMID 41567425

DOCUMENTS (1):
  • Study Protocol (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT05144724/Prot_000.pdf